CLINICAL TRIAL: NCT06476717
Title: Donor-derived Cell-free DNA (Dd-cfDNA) Monitoring to Detect Kidney Allograft Injury and Monitor the Effect Anti-rejection Treatment
Brief Title: Donor-derived Cell-free DNA in Kidney Transplant Recipients
Acronym: DEFILE
Status: Completed | Type: Observational
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Principal Investigator, Prof. Ondřej Viklický, M.D., Ph.D., Head of Department of Nephrology and Transplant Center, Institute for Clinical and Experimental Medicine
Other Study IDs: 15689/21
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-06

CONDITIONS: Kidney Transplantation; Acute Rejection of Renal Transplant
Keywords: Kidney Transplantation; Acute Rejection of Renal Transplant; dd-cfDNA; non-invasive test
MeSH Terms: interventions — Biopsy; Immunosuppression Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood samples of recipient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective monitoring within 1 year follow-up: Patients after kidney transplantation from deceased donors (n=100) were prospectively enrolled and dd-cf DNA levels were measured at defined timepoints (0, D14, 1,2,3,4,6,9 and 12 months) within 12 months.
  Interventions: Procedure: Biopsy; Diagnostic Test: Blood Biomarkers - cfDNA
- The effect of treatment cohort: Patients were enrolled at the time of biopsy with histologic and /or molecular signs of rejection. Donor-derived cell-free DNA (dd-cf DNA) were measured at the time of biopsy before centre standard of care treatment and then at weeks 1, 2 and 3 after biopsy.
  Interventions: Procedure: Biopsy; Diagnostic Test: Blood Biomarkers - cfDNA; Drug: Antirejection therapy

INTERVENTIONS:
Procedure: Biopsy — Kidney allograft biopsy
Diagnostic Test: Blood Biomarkers - cfDNA — dd-cfDNA
  Other Names: dd-cfDNA
Drug: Antirejection therapy — Patients will receive standard antirejection therapy according to center protocol.
  Groups: The effect of treatment cohort

SUMMARY:
Donor-derived cell-free DNA (dd-cfDNA) is a promising non-invasive biomarker of kidney allograft rejection. In this prospective, single center, observational monitoring study, we aim to evaluate a role of dd-cfDNA in predicting kidney allograft injuries, i.e. rejection and non-rejection injuries within 12 months, and to monitor the effect of anti rejection treatment.

DETAILED DESCRIPTION:
Kidney transplantation represents the best therapeutic option in patients with end-stage kidney disease. Among main causes of graft loss belongs kidney allograft rejection which is diagnosed based on histology/molecular assessment of biopsy sample. This is invasive procedure, but provides more precise result regarding type of rejection. Contrary, donor-derived cell-free DNA (dd-cfDNA) is a novel non-invasive biomarker of allograft rejection with excellent negative predictive power. Moreover it may be useful for predicting allograft injuries and resolution of injuries after treatment.

In the prospective cohort, 100 renal allograft patients will be enrolled and dd-cfDNA levels determined from blood collected at predefined time points (preTX, POD14, M1, 2, 3, 4, 6, 9, 12).

In the second cohort, 40 patients will be enrolled at the time of biopsy with histological and/or molecular diagnosis of rejection and dd-cfDNA levels measured just before initiation of treatment and then at week 1, 2 and 3 after biopsy.

Peripheral blood will be collected in 2x 10 ml cfDNA (Streck) collection tubes for each study visit and dd-cfDNA will be quantified by the Prospera™ test (Natera Inc., Austin, Texas).

All patients will receive standard of care treatment according to centre protocol and no patients or providers will receive the results of dd-cfDNA testing during the study. Study protocol and patient informed consent were approved by Ethical committee.

ELIGIBILITY:
Inclusion Criteria:

* Recipient age ≥ 18 years and <85 years
* Written Informed Consent cohort 1
* deceased donor kidney transplant recipient cohort 2
* patients with kidney allograft biopsy at center showing any type of rejection which is going to be treated
* patient wishing to repeatedly travel to center

Exclusion Criteria:

cohort 1

* living donor
* multiple transplant
* dual transplant
* haematopoetic stem cell transplant in a history

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients. Patients will receive standard immunosuppression based on tacrolimus, mycophenolate mofetil and steroids along with induction (basiliximab in low risk and rATG in high-risk) according to center protocol. All procedures in transplant recipients will be routine ones, included for cause biopsies and 3M protocol biopsy or antirejection therapy (standard of care in the center). Antirejection therapies are defined by center protocol and clinical team decision.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2024-05-12 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
dd-cfDNA | 12 months
  dd-cfDNA monitoring active rejection and other allograft injuries
dd-cfDNA | 4 weeks
  Monitoring of effects of antirejection treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Viklicky, M.D., Ph.D., Principal Investigator — Dept. of Nephrology, IKEM
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia, Czechia